CLINICAL TRIAL: NCT02846285
Title: Causes of Low Digestive Bleeding in Proctology
Acronym: CASPeR
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CASPeR
Record Dates: First submitted 2016-07-21; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Lower Gastrointestinal Tract; Colorectal Surgery; Proctology
Keywords: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
The various causes of bleeding Proctological are well known to gastroenterologists in clinical practice but their proportions have not, to our knowledge, been dedicated epidemiological studies. Investigators wanted to evaluate this data as part of a specialized consultation. Investigators have prospectively collected the causes of gastrointestinal bleeding down the patients seen two of us in specialized proctology center. A clinical examination including an inspection, palpation and feel, and a anoscopy (when possible) were made during the consultation. Local levies referred (s) histological and / or infection were also carried out if necessary. When she had not been made, a colonic exploration was offered to all patients over 45 years and / or when indicated by the pathological context. When there were several possible causes, the clinician holding one that seemed to be the main. Patients consulting within four months postoperatively a proctology action were not included. The study period extended from September 2013 to July 2014 inclusive. The collection of anonymous data.

DETAILED DESCRIPTION:
The various causes of bleeding Proctological are well known to gastroenterologists in clinical practice but their proportions have not, to our knowledge, been dedicated epidemiological studies. Investigators wanted to evaluate this data as part of a specialized consultation. Investigators have prospectively collected the causes of gastrointestinal bleeding down the patients seen two of us in specialized proctology center. A clinical examination including an inspection, palpation and feel, and a anoscopy (when possible) were made during the consultation. Local levies referred (s) histological and / or infection were also carried out if necessary. When she had not been made, a colonic exploration was offered to all patients over 45 years and / or when indicated by the pathological context. When there were several possible causes, the clinician holding one that seemed to be the main. Patients consulting within four months postoperatively a proctology action were not included. The study period extended from September 2013 to July 2014 inclusive. The collection of anonymous data.

ELIGIBILITY:
Inclusion Criteria:

* All patients with proctological context

Exclusion Criteria:

* Patients refusing to participate

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exploration was offered to all patients over 45 years and / or when indicated by the pathological context
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment of causes and determine the origin of down gastrointestinal bleedings | Within 4 months after surgery
  Determine the origine of gastrointestinal bleedings from the below:
  * Internal hemorrhoidal pathology
  * Anal Fissure
  * Perianal Crohn lesions
  * Cryto-glandular Anal fistula
  * Thrombosis external hemorrhoidal
  * Anal condylomata and / or perianal
  * Syndrome solitary rectal ulcer without prolapse externalized
  * Ano-radiation proctitis
  * Anal dermatitis and / or perianal
  * Complete Rectal prolapse externalized
  * Ulcerative colitis Recto
  * other

CONTACTS AND LOCATIONS:
Overall Officials: FATHALLA Nadia, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France